CLINICAL TRIAL: NCT02142647
Title: Effects of Dietary Protein From Meat vs. Dairy on Infant Growth, Body Composition and Gut Health
Brief Title: Effect of Protein From Complementary Foods on Infant Growth, Body Composition and Gut Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other); National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14-0139
Record Dates: First submitted 2014-05-14; First posted 2014-05-20 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Infant Growth; Infant Body Fat; Infant Gut Microbiome
Keywords: infant growth; dietary protein; body composition; gut microbiome
MeSH Terms: interventions — Meat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- meat group (Active Comparator): Infants in this group will receive complementary foods with high protein content mainly from meat
  Interventions: Behavioral: a high-protein complementary diet with meat
- dairy group (Active Comparator): infants in this group will receive complementary foods mainly from dairy
  Interventions: Behavioral: a high-protein complementary diet with dairy

INTERVENTIONS:
Behavioral: a high-protein complementary diet with meat — infants will consume a high-protein complementary diet with protein mainly from meat
  Arms: meat group
Behavioral: a high-protein complementary diet with dairy — infants will consume a high-protein complementary diet with protein mainly from dairy
  Arms: dairy group

SUMMARY:
Current research shows that dairy protein accelerates infant weight gain, which is a risk factor for later on obesity and metabolic syndrome. However, dietary protein from other sources haven't been studied yet. This longitudinal study will compare two complementary feeding regimens with dietary protein mainly from 1) meat; 2) dairy on infant growth, body composition and gut microbiome from 5 to 12 months of age in formula fed infants. Healthy infants at approximately 5 months of age will be randomized to either a meat protein, or a dairy protein group with complementary protein mainly from meat or dairy. Infants will consume one of these diets for 7 months (6-12 months of age) and infant growth, body composition, growth biomarkers and gut microbiome will be measured to compare between groups and over time.

DETAILED DESCRIPTION:
Two observational follow-up visits will be conducted at 18 and 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* 1-5 months of age
* Formula fed
* On breast milk less than 1 month
* Healthy
* Term Birth (36-42 weeks)
* Appropriate for gestational age

Exclusion Criteria:

* Congenital anomalies that impact feeding, growth, or development
* Low birth weight
* Not able to consume milk-based formula
* Known chronic diseases or allergies affecting protein consumption/digestion

Ages: 1 Month to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2014-03; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change of linear growth | 6 months
  growth, including linear growth (length), body weight, and all the Z scores will be recorded at the beginning and end of the study.

SECONDARY OUTCOMES:
Change in Body composition | 5 and 12 months of age
  body composition: fat mass, fat-free mass will be assessed at the beginning and end of the study

OTHER OUTCOMES:
Change in gut microbiome | 5, 9.5 and 12 months of age
  Gut microbiota profile will be measured at the beginning, mid point, and end of the intervention by collecting stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Krebs, MD, Principal Investigator — UC Denver
Locations (1):
- UC Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Odiase E, Frank DN, Young BE, Robertson CE, Kofonow JM, Davis KN, Berman LM, Krebs NF, Tang M. The Gut Microbiota Differ in Exclusively Breastfed and Formula-Fed United States Infants and are Associated with Growth Status. J Nutr. 2023 Sep;153(9):2612-2621. doi: 10.1016/j.tjnut.2023.07.009. Epub 2023 Jul 26. PMID 37506974
- [Derived] Tang M, Andersen V, Hendricks AE, Krebs NF. Different Growth Patterns Persist at 24 Months of Age in Formula-Fed Infants Randomized to Consume a Meat- or Dairy-Based Complementary Diet from 5 to 12 Months of Age. J Pediatr. 2019 Mar;206:78-82. doi: 10.1016/j.jpeds.2018.10.020. Epub 2018 Nov 6. PMID 30413312
- [Derived] Tang M, Hendricks AE, Krebs NF. A meat- or dairy-based complementary diet leads to distinct growth patterns in formula-fed infants: a randomized controlled trial. Am J Clin Nutr. 2018 May 1;107(5):734-742. doi: 10.1093/ajcn/nqy038. PMID 29722841